CLINICAL TRIAL: NCT02408250
Title: Tolerance of Early Exercise in Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0226
Record Dates: First submitted 2015-03-16; First posted 2015-04-03 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Critical Illness
Keywords: algorithm; critical illness; early exercise; feasibility; intensive care unit; physical therapy
MeSH Terms: conditions — Critical Illness; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Exercise program — Exercise program in intensive care unit established from a decisional algorithm and applied to the critical care unit patients

SUMMARY:
Practice guidelines recommend early physical therapy in intensive care unit. Feasibility, safety and efficacy are confirmed by growing evidence based data. However, the scientific literature emphasizes the heterogeneity of targeted populations, lack of precisions concerning eligibility criteria, program modalities, timing initiation, progressions and stopping criteria. However, all these results remain to be precised and confirmed. So, the investigators hypothesize that an early exercise program in intensive care unit formalized from a decisional algorithm is well tolerated in clinical practice.

DETAILED DESCRIPTION:
Practice guidelines recommend early physical therapy in intensive care unit. Feasibility, safety and efficacy are confirmed by growing evidence based data. However, the scientific literature emphasizes the heterogeneity of targeted populations, lack of precisions concerning eligibility criteria, program modalities, timing initiation, progressions and stopping criteria. However, all these results remain to be precised and confirmed. So, the investigators hypothesize that an early exercise program in intensive care unit formalized from a decisional algorithm is well tolerated in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Over 18 years old
* Hospitalized in intensive care unit
* Patients whose clinical condition allows initiating an early exercise program from critical care physician inclusion

Exclusion Criteria:

* Less than 18 years old or disabled adult
* Head or spinal severe trauma
* Severe trauma of the lower limbs or pelvis
* Musculoskeletal and neurological conditions which do not permit to realise the exercise program
* Patient for whom the reason for hospitalization does not justify early physical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critical care unit patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Score difference on a discomfort visual analogic scale between before and after program completion | at day 1

SECONDARY OUTCOMES:
Functional capacity (PFIT: Physical Function ICU Test score) | at day 1
length of stay on intensive care unit | at day 1
mortality in ICU | at day 1
Unit of discharge (specialty of the unit) | at day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France